CLINICAL TRIAL: NCT00185263
Title: A Multinational Multicenter, Randomized , Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Ad5FGF-4 in Patients With Stable Angina
Brief Title: Safety and Efficacy of Intracoronary Ad5FGF-4 in Patients With Stable Angina
Acronym: AGENT-4
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardium Therapeutics (Industry)
Responsible Party: Chief Medical Officer, Cardium Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 305602
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Stable Angina
Keywords: angina; FGF-4; angiogenesis; adenovector; growth factor; myocardial ischemia; revascularization
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Ad5FGF-4
  Interventions: Genetic: AdF5FGF-4 vs. Placebo
- 2 (Experimental): Ad5FGF-4
  Interventions: Genetic: AdF5FGF-4 vs. Placebo
- 3 (Placebo Comparator): Placebo
  Interventions: Genetic: AdF5FGF-4 vs. Placebo

INTERVENTIONS:
Genetic: AdF5FGF-4 vs. Placebo — Intracoronary infusion

SUMMARY:
The purpose of this study is to determine whether a single intracoronary infusion of Ad5FGF-4 is effective in improving exercise capacity measured by exercise treadmill testing, angina functional class, patient symptoms, quality of life, and cardiovascular outcomes. To doses are to be studied, 2.87x10(8) and 2.87x10(9) viral particles, to evaluate the dose-response of Ad5FGF-4. Short-term and long-term safety of Ad5FGF-4 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* CCS class II - IV, technically unsuitable for revascularization by CABG or PTCA able to exercise between 3 and 10 minutes on treadmill

Exclusion Criteria:

* Unstable angina, CCS class 1 angina optimal candidates for revascularization

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2002-03; Primary Completion 2005-01 (Actual); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Treadmill exercise duration | Week 12

SECONDARY OUTCOMES:
Time to coronary events | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Foster, MD, Study Director — Cardium Therapeutics, 12255 El Camino Real, Suite 250, San Diego, CA 92130, USA, +1-858-436-1000

REFERENCES:
- [Derived] Henry TD, Grines CL, Watkins MW, Dib N, Barbeau G, Moreadith R, Andrasfay T, Engler RL. Effects of Ad5FGF-4 in patients with angina: an analysis of pooled data from the AGENT-3 and AGENT-4 trials. J Am Coll Cardiol. 2007 Sep 11;50(11):1038-46. doi: 10.1016/j.jacc.2007.06.010. Epub 2007 Aug 24. PMID 17825712